CLINICAL TRIAL: NCT05992532
Title: GammaGA: Study of the Prevalence of Acid Sphingomyelinase Deficiency Disease (ASMD) and Gaucher Disease in Patients With Monoclonal Gammopathies and/or Multiple Myeloma
Brief Title: GammaGA: Prevalence of Acid Sphingomyelinase Deficiency Disease (ASMD) and Gaucher Disease in Patients With Monoclonal Gammopathies and/or Multiple Myeloma
Status: Recruiting | Type: Observational
Sponsor: Fundación Española de Hematología y Hemoterapía (Other)
Responsible Party: Sponsor
Other Study IDs: GammaGA
Record Dates: First submitted 2023-08-08; First posted 2023-08-15 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Gaucher Disease; Acid SphingoMyelinase Deficiency
Keywords: Gaucher disease; Acid sphingomyelinase deficiency; GD; ASMD; DBS; Splenomegaly; monoclonal gammopathies; multiple myeloma
MeSH Terms: conditions — Gaucher Disease; Niemann-Pick Diseases; Splenomegaly; Paraproteinemias; Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study of splenomegaly, and the follow-up of splenectomized patients, is one of the causes of referral of these patients to pediatric gastroenterology and oncohematology clinics, and adult internal medicine and hematology. The study and management of splenomegaly is well described among the different medical specialties to which these patients arrive. After the application of the different algorithms and the different studies that are carried out, these splenomegaly are identified as being of hepatic, infectious, inflammatory, congestive, hematological origin and primary causes. Despite these studies of splenomegaly, approximately 10-15% of these patients still remain undiagnosed.

Several studies have suggested that there is an increased frequency of MGUS (monoclonal gammopathy of undetermined significance) and/or multiple myeloma (MM) among Gaucher patients. Regarding ASMD (Acid Sphingomyelinase Deficiency), few studies have been published but it seems the 21% of patient with ASMD has MGUS and 15% ASMD patients have MGUS. Moreover, patients with MGUS and Gaucher disease (GD) are at increased risk of developing MM.

The objective of the present study is to increase the diagnostic sensitivity of these unknown splenomegalys, or unknown splenomegaly patients with MGUS or multiple myeoloma who remain in consultations, using the usual diagnostic clinical procedures of unknown splenomegaly and unknown splenectomy patients, where we include the extraction of a blood sample for dry drop test (DBS), where the determination of the enzymatic/genetic activity will be carried out for Gaucher disease (GD) and acid sphingomyelinase deficiency (ASMD) , analysis of LisoGl1 and LisoSM.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients of both sexes.
* Patients with splenomegaly (spleen palpable at ≥ 1cm from the costal margin) or splenectomy not related to any specific condition, or patients with thrombocytopenia (with or without splenomegaly). In cases where the patient is undergoing treatment for their underlying condition, the thrombocytopenia must have been present prior to the start of the treatment.
* Patient who gives their consent to participate in the study.

Exclusion Criteria:

* Splenomegaly due to portal hypertension (documented by abdominal ultrasound or other instrumental test) due to liver disease
* Hematologic malignancy [documented by positive physical exam + blood smear or fine needle aspiration (FNA) or bone marrow biopsy]
* Hemolytic anemia and/or thalassemia
* Patients who cannot meet the requirements of the protocol due to mental and/or cognitive alterations, uncooperative patients, educational limitations and understanding of written language
* Refusal of the patient to participate in the study

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Adult patients of both sexes.
  * Patients who present signs, assessed instrumentally or with laboratory tests, of unknown splenomegaly, defined as a palpable spleen ≥ 1cm from the costal margin or diagnosed by ultrasound, magnetic resonance imaging (MRI) or computed tomography (CT) of the spleen.
  * Splenectomy patient with no diagnosis of the origin of the splenomegaly of unknown origin.
  * Patients with thrombocytopenia. In cases where the patient is undergoing treatment for their underlying condition, the thrombocytopenia must have been present prior to the start of the treatment
Sampling Method: Non-Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2023-05-30 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Gaucher disease (GD) and acid sphingomyelinase deficiency (ASMD) | 36 months
  Determinate the prevalence of Gaucher disease (GD) and acid sphingomyelinase deficiency (ASMD)

CONTACTS AND LOCATIONS:
Locations (23):
- Spain (23):
  - Hospital Universitario de Álava, Vitoria-Gasteiz, Alava
  - Hospital Universitario Torrecárdenas, Almería, Almería
  - Hospital Son Espases, Palma de Mallorca, Balearic Islands
  - Hospital Parc Taulí, Sabadell, Barcelona
  - Hospital Universitario de Burgos, Burgos, Burgos
  - Hospital de Valdepeñas, Valdepeñas, Ciudad Real
  - Hospital Universitario Dr. Josep Trueta, Girona, Girona
  - Hospital Universitario Virgen de las Nieves, Granada, Granada
  - Hospital San Jorge, Huesca, Huesca
  - Hospital de Jaén, Jaén, Jaén
  - Hospital del Bierzo, Ponferrada, León
  - Hospital Arnau de Vilanova, Lleida, Lleida
  - Hospital Universitario La Paz, Madrid, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid, Madrid
  - Hospital Fundación Jiménez Díaz, Madrid, Madrid
  - Hospital Regional Universitario de Málaga, Málaga, Málaga
  - Complejo Hospitalario Universitario de Orense, Ourense, Orense
  - Hospital Alvaro Cunqueiro, Vigo, Pontevedra
  - Hospital Alcañiz, Alcañiz, Teruel
  - Hospital de Manises, Valencia, Valencia
  - Hospital Universitario y Politécnico La Fe, Valencia, Valencia
  - Hospital Clínico Universitario de Valladolid, Valladolid, Zaragoza
  - Complejo Asistencial de Ávila, Ávila, Ávila